CLINICAL TRIAL: NCT04847232
Title: An International, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Sodium Zirconium Cyclosilicate on Arrythmia-related Cardiovascular Outcomes in Participants on Chronic Hemodialysis With Recurrent Hyperkalemia (DIALIZE-Outcomes)
Brief Title: Effect of Sodium Zirconium Cyclosilicate on Arrythmia-related Cardiovascular Outcomes in Participants on Chronic Hemodialysis With Recurrent Hyperkalemia (DIALIZE-Outcomes)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The event rate observed in the study continued to be below primary assumptions, so that the completion of the study within a reasonable timeframe was deemed very unlikely.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9487C00001; 2020-005561-14 (EudraCT Number)
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hyperkalemia
Keywords: Hemodialysis; Hyperkalemia; Cardiovascular Events; Atrial Fibrillation; Ventricular Tachycardia
MeSH Terms: conditions — Hyperkalemia; Atrial Fibrillation; Tachycardia, Ventricular | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sodium Zirconium Cyclosilicate (Experimental)
  Interventions: Drug: Sodium Zirconium Cyclosilicate (SZC)
- Placebo (Placebo Comparator)
  Interventions: Drug: SZC Placebo

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate (SZC) — Powder for oral suspension in a sachet. A dose is titrated in 5 g increments during a period of 4 weeks from 5 g up to 15 g qd on non-dialysis days. Afterward, the dose is adjusted monthly (or more frequent based on clinical judgment) depending on the current potassium value as measured after the long interdialytic interval (LIDI).
  Other Names: Lokelma TM
  Arms: Sodium Zirconium Cyclosilicate
Drug: SZC Placebo — Powder for oral suspension in a sachet. A dose is titrated in 5 g increments during a period of 4 weeks from 5 g up to 15 g qd on non-dialysis days. Afterward, the dose is adjusted monthly (or more frequent based on clinical judgment) depending on the current potassium value as measured after the LIDI.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of Sodium Zirconium Cyclosilicate (SZC) on arrhythmia-related cardiovascular outcomes in participants on chronic hemodialysis with recurrent hyperkalemia.

DETAILED DESCRIPTION:
This is an international, multicenter, event-driven, randomized, double-blind, parallel group, placebo-controlled study, evaluating the utility of SZC versus placebo to reduce the incidence of sudden cardiac death (SCD), stroke, and arrhythmia-related hospitalizations, interventions, and emergency department (ED) visits in participants on chronic hemodialysis with recurrent hyperkalemia.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol
2. Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses
3. Must be ≥ 18 years of age, at the time of signing the ICF.
4. Receiving hemodialysis (or hemodiafiltration) 3 times a week for treatment of ESRD for ≥ 4 months before enrollment
5. Must have hemodialysis access consisting of an arteriovenous fistula, arteriovenous graft, or tunneled (permanent) catheter which is expected to remain in place for the entire duration of the study
6. At least 2 out of 3 pre-dialysis S K ≥ 5.5 mmol/L after the LIDI during screening
7. Negative pregnancy test for female participants of childbearing potential
8. Female participants must be 1 year postmenopausal, surgically sterile, or using one highly effective form of birth control (defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly). They should have been stable on their chosen method of birth control for a minimum of 3 months before entering the study and willing to remain on the birth control until 12 weeks after the last dose

Exclusion Criteria:

1. Pseudohyperkalemia secondary to hemolyzed blood specimen (this situation is not considered screening failure, sampling or full screening can be postponed to a later time as applicable)
2. Presence of cardiac arrhythmias or conduction defects that require immediate treatment
3. Participants who have a pacemaker or implantable cardiac defibrillator
4. Any medical condition, including active, clinically significant infection or liver disease, that in the opinion of the investigator or sponsor may pose a safety risk to a participant in this study, confound safety or efficacy assessment and jeopardize the quality of the data, or interfere with study participation, or any other restrictions or contraindications in the local prescribing information for SZC
5. History of QT prolongation associated with other medications that required discontinuation of that medication
6. Congenital long QT syndrome
7. QTcF > 550 msec
8. Atrial fibrillation requiring immediate/urgent intervention at screening or randomizations
9. Treated with sodium polystyrene sulfonate (SPS, Kayexalate, Resonium), calcium polystyrene sulfonate (CPS Resonium Calcium), patiromer (Veltassa), or SZC (Lokelma) within 7 days before screening or anticipated requiring chronic use of any of these agents during the study. If participant requires rescue therapy (potassium binder or dialysate S-K change during screening period), the participant will be screen failed
10. Participation in another clinical study with an investigational product, device, or non-standard hemodialysis procedure administered within one month before screening
11. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
12. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements
13. Previous randomization in the present study
14. Females who are pregnant (confirmed with positive pregnancy test or a uterine ultrasound if pregnancy test result is questionable), breastfeeding, or planning to become pregnant during the study
15. Known hypersensitivity or previous anaphylaxis to SZC or to components thereof
16. Scheduled date for living donor kidney transplant
17. Sustained Ventricular Tachycardia > 30 seconds requiring assessment / intervention

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2690 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fishbane, Professor, MD, Principal Investigator — North Shore University Hospital, 300 Community Drive, Manhasset, NY 11030
Locations (288):
- United States (50):
  - Research Site, Huntsville, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Glendale, California
  - Research Site, Granada Hills, California
  - Research Site, Lynwood, California
  - Research Site, San Diego, California
  - Research Site, Vacaville, California
  - Research Site, Victorville, California
  - Research Site, Denver, Colorado
  - Research Site, Bloomfield, Connecticut
  - Research Site, Middlebury, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Tampa, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Statesboro, Georgia
  - Research Site, Nampa, Idaho
  - Research Site, Iowa City, Iowa
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Roseville, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Brookhaven, Mississippi
  - Research Site, Columbus, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Jersey City, New Jersey
  - Research Site, Manhasset, New York
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Spartanburg, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Conroe, Texas
  - Research Site, El Paso, Texas
  - Research Site, Greenville, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, St. George, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (7):
  - Research Site, Córdoba
  - Research Site, Junín
  - Research Site, Mar del Plata
  - Research Site, Pergamino
  - Research Site, San Luis
  - Research Site, Santa Rosa
  - Research Site, Sarandí
- Austria (2):
  - Research Site, Graz
  - Research Site, Innsbruck
- Brazil (9):
  - Research Site, Brasília
  - Research Site, Curitiba
  - Research Site, Joinville
  - Research Site, Maringá
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (14):
  - Research Site, Blagoevgrad
  - Research Site, Gotse Delchev
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Razlog
  - Research Site, Samokov
  - Research Site, Sandanski
  - Research Site, Silistra
  - Research Site, Smolyan
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Yambol
- Canada (8):
  - Research Site, Saint John, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (46):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Dongguan
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guilin
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Huai'an
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Jiujiang
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanyang
  - Research Site, Ningbo
  - Research Site, Panjin
  - Research Site, Pingxiang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Shenzhen
  - Research Site, Siping
  - Research Site, Taian
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuhu
  - Research Site, Wuxi
  - Research Site, Xiamen
  - Research Site, Xianyang
  - Research Site, Yibin
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
  - Research Site, Zhuzhou
- Czechia (10):
  - Research Site, České Budějovice
  - Research Site, Havlíčkův Brod
  - Research Site, Jilemnice
  - Research Site, Klatovy
  - Research Site, Liberec
  - Research Site, Nové Město na Moravě
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Tábor
  - Research Site, Třebíč
- Germany (7):
  - Research Site, Cloppenburg
  - Research Site, Düsseldorf
  - Research Site, Hanover
  - Research Site, Minden
  - Research Site, Potsdam
  - Research Site, Stuttgart
  - Research Site, Villingen-Schwenningen
- Hungary (8):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Kaposvár
  - Research Site, Karcag
  - Research Site, Kistarcsa
  - Research Site, Miskolc
  - Research Site, Nagykanizsa
  - Research Site, Szombathely
- India (5):
  - Research Site, Ahmedabad
  - Research Site, Chennai
  - Research Site, Dhanvantari Nagar
  - Research Site, Nadiād
  - Research Site, Pune
- Italy (12):
  - Research Site, Bassano del Grappa
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Caserta
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Pesaro
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo
  - Research Site, Verona
- Japan (22):
  - Research Site, Fujisawa-shi
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Kawasaki-shi
  - Research Site, Kumagaya-shi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Moriya-shi
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nakagami-gun
  - Research Site, Okinawa-shi
  - Research Site, Ōmihachiman
  - Research Site, Sashima-gun
  - Research Site, Setagaya-ku
  - Research Site, Shiroishi-shi
  - Research Site, Tamanashi
  - Research Site, Toride-shi
  - Research Site, Tsuchiura-shi
  - Research Site, Tsukuba
  - Research Site, Ushiku-shi
  - Research Site, Yatomi-shi
- Malaysia (4):
  - Research Site, Batu Caves
  - Research Site, Ipoh
  - Research Site, Malacca
  - Research Site, Seri Manjung
- Mexico (11):
  - Research Site, Chihuahua City
  - Research Site, Culiacán
  - Research Site, D.F
  - Research Site, Mazatlán
  - Research Site, Mexico City
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, San Luis Potosí City
  - Research Site, Veracruz
  - Research Site, Xalapa
  - Research Site, Zapopan
- Peru (3):
  - Research Site, Cusco
  - Research Site, Lima
  - Research Site, Piura
- Poland (13):
  - Research Site, Gdansk
  - Research Site, Leżajsk
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Oleśnica
  - Research Site, Olkusz
  - Research Site, Pszczyna
  - Research Site, Słupsk
  - Research Site, Tczew
  - Research Site, Wołomin
  - Research Site, Wroclaw
  - Research Site, Żory
  - Research Site, Żyrardów
- Russia (7):
  - Research Site, Kemerovo
  - Research Site, Mytischi
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Penza
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Slovakia (6):
  - Research Site, Bratislava
  - Research Site, Komárno
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Púchov
  - Research Site, Žilina
- Spain (6):
  - Research Site, Alcalá de Henares
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Valencia
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, Linkou District
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Ratchathewi
- Turkey (Türkiye) (6):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Gaziantep
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
- Ukraine (9):
  - Research Site, Chernivtsі
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- United Kingdom (8):
  - Research Site, Bristol
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Preston
  - Research Site, Salford
  - Research Site, Swansea
  - Research Site, Wolverhampton
- Vietnam (5):
  - Research Site, Biên Hòa
  - Research Site, Da Nang
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Fishbane S, Dember LM, Jadoul M, Kovesdy CP, Guzman N, Kordzakhia G, Lisovskaja V, Sekar P, Wessman P, Al-Shurbaji A, Herzog CA. The randomized DIALIZE-Outcomes trial evaluated sodium zirconium cyclosilicate in hemodialysis. Kidney Int. 2025 Oct;108(4):686-694. doi: 10.1016/j.kint.2025.06.016. Epub 2025 Jul 4. PMID 40618849
- [Derived] Fishbane S, Jadoul M, Dember L, Kovesdy CP, Al-Shurbaji A, Lisovskaja V, Sekar P, Katona B, Guzman N, Herzog C. Evaluation of the effect of sodium zirconium cyclosilicate on arrhythmia-related cardiovascular outcomes in patients receiving chronic haemodialysis with hyperkalaemia: protocol for the multicentre, randomised, controlled DIALIZE-Outcomes study. BMJ Open. 2023 May 25;13(5):e071309. doi: 10.1136/bmjopen-2022-071309. PMID 37230521
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9487C00001&attachmentIdentifier=7bd2ebb1-fd15-4ffd-b33a-18d3d5a2dca1&fileName=D9487C00001_-_Redacted_CSP.pdf&versionIdentifier=
- See also: Statistical Analysis Plan - Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9487C00001&attachmentIdentifier=ad595187-fc73-4fb0-9926-63b53fddc652&fileName=D9487C00001_-_Statistical_Analysis_Plan_-_Redacted.pdf&versionIdentifier=
- See also: D9487C00001_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9487C00001&attachmentIdentifier=a726e622-6a0f-4d71-b0f7-711400766969&fileName=D9487C00001_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- SZC (Active): 5 g SZC QD to 15 g SZC QD
- Placebo: SZC Placebo
Period: Overall Study
Arm/Group | SZC (Active) | Placebo
Started | 1349 | 1341
Completed | 0 | 0
Not Completed | 1349 | 1341
Not completed — Death | 123 | 115
Not completed — Lost to Follow-up | 3 | 10
Not completed — Withdrawal by Subject | 73 | 101
Not completed — Subcategories under "Other" not reported. | 1150 | 1115

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SZC (Active) | Placebo | Total
Number analyzed (Participants) | 1349 | 1341 | 2690
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.8 (13.3) | 56.3 (13.6) | 56.1 (13.4)
Age, Customized [Number; unit: Participants]
  18 yr ≤ Age < 51 yr | 442 | 441 | 883
  51 yr ≤ Age < 65 yr | 526 | 509 | 1035
  65 yr ≤ Age < 85 yr | 373 | 378 | 751
  Age ≥ 85 yr | 8 | 13 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 498 | 517 | 1015
  Male | 851 | 824 | 1675
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 49 | 52 | 101
  ASIAN | 392 | 389 | 781
  BLACK OR AFRICAN AMERICAN | 121 | 130 | 251
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 3 | 2 | 5
  WHITE | 688 | 672 | 1360
  OTHER | 75 | 86 | 161
  NOT REPORTED | 21 | 10 | 31
spKt/V [Mean (Standard Deviation); unit: Dimensionless] — Dialysis adequacy, single-pool Kt/V. The parameter Kt/V is a measurement of the efficacy of a hemodialysis session. It identifies the effective removal of a specific solute (clearance K) resulting from a given treatment (characterized by time t) in each patient (with a specific volume of distribution V for the solute considered). Operationally, Kt/V is a dimensionless number. Population: Full analysis set; participants with a non-missing value.
  Dimensionless
    number analyzed (Participants) | 1007 | 994 | 2001
    (all) | 1.48 (0.39) | 1.51 (0.47) | 1.49 (0.43)
Dialysis vintage [Mean (Standard Deviation); unit: Years] — Time since first dialysis. Population: Full analysis set; participants with a non-missing value.
  Years
    number analyzed (Participants) | 1349 | 1337 | 2686
    (all) | 6.01 (5.41) | 5.82 (5.20) | 5.92 (5.31)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of the Composite of Cardiac Event Outcomes
Description: Incidence of the composite endpoint of SCD, all stroke, or hospitalization/intervention/emergency department (ED) visit due to arrhythmias is analyzed based on Cox regression model with treatment and region as covariates. Patients with no events are censored at final clinical assessment, death, or disposition event.
Time Frame: From Randomization (Visit 4) up to week 129 (Randomized Study Intervention Phase)
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | SZC (Active) | Placebo
Number analyzed (Participants) | 1349 | 1341
Participants | 119 | 119
Statistical Analysis 1: Comparison: SZC (Active) vs Placebo; Test type: Other — Test of HR = 1; p = 0.867, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.76 to 1.26] — SZC relative to Placebo

2. Secondary Outcome: Normokalemia at 12 Months Post-randomization
Description: Logistic regression analysis of whether a subject is Normokalemic (S-K of 4.0 - 5.5 mmol/L ) after the LIDI at the 12-month visit.
Time Frame: Randomization to 12-Month Visit
Population: Full analysis set. Only subjects with non-missing S-K value at the 12 month visit included in the analysis.
Measure: Number; unit: Participants with event
Arm/Group | SZC (Active) | Placebo
Number analyzed (Participants) | 669 | 624
Participants with event | 495 | 293
Statistical Analysis 1: Comparison: SZC (Active) vs Placebo; Test type: Other — Test of OR = 1; p < .0001, Regression, Logistic; Odds Ratio (OR) = 3.36, 95% CI 2-sided [2.64 to 4.26] — SZC relative to Placebo

3. Secondary Outcome: Incidence of the Composite of Arrhythmia Related Events
Description: Incidence of the composite endpoint of hospitalization, intervention, emergency department (ED) visit due to arrhythmias is analyzed based on Cox regression model with treatment and region as covariates. Patients with no events are censored at final clinical assessment, death, or disposition event.
Time Frame: From Randomization (Visit 4) up to week 129 (Randomized Study Intervention Phase)
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | SZC (Active) | Placebo
Number analyzed (Participants) | 1349 | 1341
Participants | 74 | 65
Statistical Analysis 1: Comparison: SZC (Active) vs Placebo; Test type: Other — Test of HR = 1; p = 0.510, Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.80 to 1.56] — SZC relative to Placebo

ADVERSE EVENTS:
Time Frame: From Randomization (Visit 4) up to week 129 (Randomized Study Intervention Phase)
Arm/Group | SZC (Active) | Placebo
All-Cause Mortality (participants affected / at risk) | 120/1348 | 113/1338
Serious Adverse Events (participants affected / at risk) | 521/1348 | 503/1338
Other Adverse Events (participants affected / at risk) | 558/1348 | 616/1338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SZC (Active) (N=1348) | Placebo (N=1338)
Acute myocardial infarction (Cardiac disorders) | 26 (30) | 19 (21)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 2 (3)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 4 (4)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 8 (8) | 5 (5)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Angina unstable (Cardiac disorders) | 3 (4) | 8 (8)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 2 (3)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Periodontal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Accidental death (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (4) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 3 (3)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 15 (15) | 12 (12)
Arrhythmia (Cardiac disorders) | 3 (3) | 1 (1)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 2 (2)
Medical device site haemorrhage (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 2 (2)
Necrosis (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 4 (5) | 3 (3)
Prosthetic cardiac valve thrombosis (General disorders) | 0 (0) | 1 (1)
Puncture site pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Sudden cardiac death (General disorders) | 9 (9) | 12 (12)
Sudden death (General disorders) | 4 (4) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 3 (4)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 15 (21) | 14 (15)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 4 (4) | 3 (3)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 2 (2)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 3 (3) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 5 (5) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 2 (3) | 2 (2)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacillus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 5 (5) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 2 (2) | 0 (0)
Bone tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 5 (5)
Covid-19 (Infections and infestations) | 19 (19) | 16 (16)
Covid-19 pneumonia (Infections and infestations) | 21 (22) | 20 (21)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 4 (4)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 12 (12) | 4 (4)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 3 (3) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 12 (16) | 8 (13)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 1 (1)
Device related bacteraemia (Infections and infestations) | 3 (3) | 3 (4)
Device related infection (Infections and infestations) | 9 (11) | 6 (6)
Device related sepsis (Infections and infestations) | 5 (5) | 2 (2)
Diabetic foot infection (Infections and infestations) | 2 (2) | 1 (1)
Diabetic gangrene (Infections and infestations) | 2 (2) | 2 (3)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 2 (2)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (3)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 9 (12) | 2 (2)
Gas gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 3 (3)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Haematological infection (Infections and infestations) | 2 (2) | 3 (3)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter duodenitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis c (Infections and infestations) | 0 (0) | 1 (1)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 4 (4)
Cardiac arrest (Cardiac disorders) | 14 (15) | 11 (11)
Infectious pleural effusion (Infections and infestations) | 2 (2) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 5 (5) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Latent tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 4 (5) | 4 (4)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0)
Ludwig angina (Infections and infestations) | 0 (0) | 1 (1)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 4 (4) | 7 (7)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 61 (75) | 60 (69)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 2 (2) | 2 (2)
Post procedural infection (Infections and infestations) | 0 (0) | 2 (2)
Post-acute covid-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Cardiac dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 3 (3)
Pyonephrosis (Infections and infestations) | 0 (0) | 1 (1)
Renal graft infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Sepsis (Infections and infestations) | 36 (38) | 20 (22)
Septic shock (Infections and infestations) | 11 (14) | 13 (13)
Shunt infection (Infections and infestations) | 0 (0) | 1 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (2)
Spontaneous bacterial peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 12 (13) | 8 (8)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 3 (3)
Staphylococcal infection (Infections and infestations) | 2 (3) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 5 (5)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0)
Suspected covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (7) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 7 (8) | 11 (12)
Urosepsis (Infections and infestations) | 0 (0) | 4 (4)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula maturation failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 11 (15) | 17 (18)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 3 (3) | 2 (2)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Arteriovenous fistula site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 16 (22) | 21 (22)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 6 (11)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fat embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 3 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Kidney rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 4 (4)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Shunt aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Shunt occlusion (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 4 (4)
Shunt stenosis (Injury, poisoning and procedural complications) | 3 (6) | 7 (16)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tracheal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electrocardiogram pr prolongation (Investigations) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Electrocardiogram qrs complex prolonged (Investigations) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Calciphylaxis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4) | 5 (5)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperglycaemic crisis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 15 (19) | 39 (56)
Hypervolaemia (Metabolism and nutrition disorders) | 22 (26) | 16 (20)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
High turnover osteopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (3)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 5 (5) | 3 (4)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 3 (3)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Cerebellar ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 3 (3)
Cerebral infarction (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 3 (3)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 5 (5) | 2 (2)
Epilepsy (Nervous system disorders) | 3 (3) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 7 (8) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypocalcaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 3 (3)
Ischaemic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 6 (6) | 14 (14)
Lacunar infarction (Nervous system disorders) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Middle cerebral artery stroke (Nervous system disorders) | 1 (1) | 1 (1)
Neurodegenerative disorder (Nervous system disorders) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Pericarditis uraemic (Cardiac disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Psychogenic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Putamen haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 4 (4) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 2 (2)
Device breakage (Product Issues) | 1 (1) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 6 (6) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Prosthetic cardiac valve failure (Product Issues) | 0 (0) | 1 (1)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Emotional distress (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 4 (4) | 3 (3)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst ruptured (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal haematoma (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 2 (2) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Noninfective oophoritis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (11)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 11 (13)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (7)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (4)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 3 (4)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (3) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Assisted suicide (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2) | 2 (2)
Aortitis (Vascular disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Diabetic macroangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dialysis hypotension (Vascular disorders) | 1 (1) | 3 (3)
Dialysis induced hypertension (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1) | 1 (1)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 3 (3)
Haematoma (Vascular disorders) | 2 (2) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 10 (12) | 8 (9)
Hypertensive crisis (Vascular disorders) | 3 (3) | 8 (10)
Hypertensive emergency (Vascular disorders) | 9 (9) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 3 (3) | 4 (5)
Hypotension (Vascular disorders) | 8 (8) | 4 (4)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 7 (8) | 9 (9)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Hyperadrenocorticism (Endocrine disorders) | 1 (1) | 0 (0)
Peripheral vein stenosis (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Polyarteritis nodosa (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein stenosis (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Vascular insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 2 (2) | 3 (3)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous occlusion (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Hyperparathyroidism tertiary (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thyrotoxic crisis (Endocrine disorders) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 5 (5) | 3 (3)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (3) | 3 (3)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 4 (5)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 2 (3) | 1 (1)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 (11) | 10 (10)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SZC (Active) (N=1348) | Placebo (N=1338)
Nausea (Gastrointestinal disorders) | 43 (51) | 59 (66)
Vomiting (Gastrointestinal disorders) | 44 (49) | 54 (69)
Pyrexia (General disorders) | 50 (59) | 45 (62)
Covid-19 (Infections and infestations) | 145 (153) | 122 (126)
Anaemia (Blood and lymphatic system disorders) | 64 (85) | 44 (55)
Pneumonia (Infections and infestations) | 50 (55) | 30 (33)
Upper respiratory tract infection (Infections and infestations) | 39 (56) | 52 (59)
Hyperkalaemia (Metabolism and nutrition disorders) | 125 (188) | 280 (480)
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 (59) | 54 (62)
Back pain (Musculoskeletal and connective tissue disorders) | 43 (50) | 25 (31)
Headache (Nervous system disorders) | 48 (63) | 52 (71)
Cough (Respiratory, thoracic and mediastinal disorders) | 47 (52) | 41 (52)
Dialysis hypotension (Vascular disorders) | 55 (170) | 59 (239)
Hypertension (Vascular disorders) | 80 (180) | 82 (171)
Constipation (Gastrointestinal disorders) | 76 (94) | 57 (74)
Diarrhoea (Gastrointestinal disorders) | 98 (122) | 93 (117)

LIMITATIONS AND CAVEATS:
Study was terminated early due to lower-than-expected primary event rate and higher than anticipated drop-out rate. Lower number of evaluable events reduces the precision of the primary analysis considerably.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT04847232/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT04847232/SAP_001.pdf